CLINICAL TRIAL: NCT04633954
Title: The Effect if Brimonidine 0.15% on the Development of Subconjunctival Hemorrhage Following Femtosecond Laser Assisted Cataract Surgery
Brief Title: Brimonidine for Subconjunctival Hemorrhage From Femtosecond Laser Assisted Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uptown Eye Specialists (Other)
Responsible Party: Principal Investigator, Sohel Somani, Ophthalmologist & Medical Director, Uptown Eye Specialists
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Red Eye 1.0
Record Dates: First submitted 2020-11-08; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Subconjunctival Hemorrhage; Cataract Surgery
Keywords: Brimonidine Tartrate; Femtosecond laser assisted cataract surgery; Bulbar redness; Subconjunctival hemorrhage; Cataract Surgery
MeSH Terms: interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brimonidine Group (Experimental): Patients in this arm receive an extra drop of brimonidine in addition to routine eye drops prior to femtosecond laser assisted cataract surgery (FLACS)
  Interventions: Drug: Brimonidine Tartrate 0.15% Oph Soln
- Control Group (No Intervention): Patients in this arm only receive routine eye drops prior to femtosecond laser assisted cataract surgery (FLACS)

INTERVENTIONS:
Drug: Brimonidine Tartrate 0.15% Oph Soln — One drop of Brimonidine Tartrate 0.15% Oph Soln prior to FLACS
  Arms: Brimonidine Group

SUMMARY:
Laser-assisted cataract surgery is a common and precise procedure done to remove cataracts from the eye. This procedure involves putting on a suction cup that applies a mild vacuum seal around the eye to stabilize the eye during the laser procedure. This suction cup often causes some bleeding under the conjunctiva around the eye which takes a few days to disappear.

The purpose of this study is to test the use of a well-known eye medication (normally for treating glaucoma) called Brimonidine tartrate 0.15% (or Alphagan-P) in patients having laser-assisted cataract surgery. The use of Brimonidine to reduce bleeding under the conjunctiva is investigational, which means it has not been approved by Health Canada for use outside of research studies like this one.

This study will see if Brimonidine will help to reduce bleeding under the conjunctiva in patients having laser-assisted cataract surgery.

DETAILED DESCRIPTION:
The focus of this study is to assess how the quality of care for patients undergoing Femtosecond laser-assisted cataract surgery (FLACS) can be improved through the application of Brimonidine Tartrate 0.15% prior to the surgery. The surgery consists of the application of a vacuum which can result in subconjunctival hemorrhage, a benign disorder. The importance of this study is due to the considerable alarm and anxiety caused to the patients by the hemorrhage which may cause them to seek our further unnecessary medical help and reduce their ability to return to work or productivity.

During the laser component of FLACS, the operated eye is secured with a suction cup or ring with vacuum that causes significant subconjunctival hemorrhage. Brimonidine is a selective alpha-2-adrenergic agonist that is a commonly used as a topical medication to treat glaucoma. Besides its intraocular pressure lowering effect, it also has a vasoconstrictive effect. This latter effect has been exploited to reduce bleeding in LASIK, cataract surgery, strabismus surgery, as well as intravitreal injections. This study will examine the effectiveness of Brimonidine to reduce subconjunctival hemorrhage during Femtosecond laser-assisted cataract surgery.

Potential side effects of topical application of Brimonidine eye drop may include blurred or loss of vision, burning, dry, or itching eyes, discharge or excessive tearing, disturbed color perception, double vision, halos around lights, headache, itching of the eye, night blindness, overbright appearance of lights, redness of the eye or inner lining of the eyelid, swelling of the eyelid, tearing of the eye, tunnel vision. The risk of this study to the subject is negligible.

To evaluate the degree of subconjunctival hemorrhage occurring in subjects undergoing Femtosecond laser-assisted cataract surgery, following preoperative application of Brimonidine 0.15%. Subconjunctival hemorrhage and its associated bulbar redness will be measured using Bulbar Redness Score using the Oculus M5 following the surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are schedules for femtosecond laser assisted cataract surgery who have provided informed consent, in accordance with application regulations and guidelines

Exclusion Criteria:

* Patients who have been on anticoagulation or antiplatelet therapy
* Patients who have undergone any conjunctival surgery in the past
* Any complication during cataract extraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Bulbar Redness Score | Pre-operatively
  Bulbar redness score measured with Oculus 5M Keratograph will detect the amount of redness before and after FLACS. The Oculus Keratograph 5M BR score uses a clinical grading scale of 0.0-4.0 in 0.1 step. A higher score correlates to increased bulbar redness.
Bulbar Redness Score | 15 minutes post-operatively
  Bulbar redness score measured with Oculus 5M Keratograph will detect the amount of redness before and after FLACS. The Oculus Keratograph 5M BR score uses a clinical grading scale of 0.0-4.0 in 0.1 step. A higher score correlates to increased bulbar redness.

SECONDARY OUTCOMES:
Analyzed Area | Pre-operatively
  Bulbar redness scoring by Oculus 5M Keratograph imaging simultaneously calculates the area analyzed, which will be compared between groups to ensure a similar surface area is measured.
Analyzed Area | 15 minutes post-operatively
  Bulbar redness scoring by Oculus 5M Keratograph imaging simultaneously calculates the area analyzed, which will be compared between groups to ensure a similar surface area is measured.
Attempts of Vacuum | During the operation
  The number of attempts it takes to achieve adequate vacuum as part of FLACS will be recorded
Duration of surgery | During the operation
  The entire duration (start to end) of the surgery will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Uptown Eye Speicialists, Brampton, Ontario, Canada

REFERENCES:
- [Background] Pasquali TA, Aufderheide A, Brinton JP, Avila MR, Stahl ED, Durrie DS. Dilute brimonidine to improve patient comfort and subconjunctival hemorrhage after LASIK. J Refract Surg. 2013 Jul;29(7):469-75. doi: 10.3928/1081597X-20130617-05. PMID 23820229
- [Background] Kim CS, Nam KY, Kim JY. Effect of prophylactic topical brimonidine (0.15%) administration on the development of subconjunctival hemorrhage after intravitreal injection. Retina. 2011 Feb;31(2):389-92. doi: 10.1097/IAE.0b013e3181eef28e. PMID 20890238
- [Background] Norden RA. Effect of prophylactic brimonidine on bleeding complications and flap adherence after laser in situ keratomileusis. J Refract Surg. 2002 Jul-Aug;18(4):468-71. doi: 10.3928/1081-597X-20020701-10. PMID 12160159
- [Background] Desco MC, Navea A, Ferrer E, Menezo JL. Effect of prophylactic brimonidine on bleeding complications after cataract surgery. Eur J Ophthalmol. 2005 Mar-Apr;15(2):228-32. doi: 10.1177/112067210501500209. PMID 15812765
- [Background] Hong S, Kim CY, Seong GJ, Han SH. Effect of prophylactic brimonidine instillation on bleeding during strabismus surgery in adults. Am J Ophthalmol. 2007 Sep;144(3):469-70. doi: 10.1016/j.ajo.2007.04.038. PMID 17765438